CLINICAL TRIAL: NCT03990701
Title: Primary Aldosteronism and Surgically Curable Forms in Hypertension Patients Using 11C-Metomidate
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: National University Health System, Singapore (Other); Clinical Imaging Research Centre (Unknown); Singapore General Hospital (Other); Tan Tock Seng Hospital (Other); Khoo Teck Puat Hospital (Other); Ng Teng Fong General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA_CURE
Record Dates: First submitted 2018-12-19; First posted 2019-06-19 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Primary Aldosteronism; Primary Aldosteronism Due to Aldosterone Producing Adenoma
Keywords: 11-C Metomidate PET/CT; Hypertension; Adrenalectomy; Adrenal Vein Sampling; Subtyping
MeSH Terms: conditions — Hyperaldosteronism; Hypertension

STUDY DESIGN:
Intervention Model Description: 11C-metomidate will be manufactured in Clinical Imaging Research Centre in compliance with good manufacturing practice using a General Electric Medical Systems PET trace 860 cyclotron. Non-contrast CT images will be acquired over the adrenal. After an intravenous injection of 11C-metomidate, PET images will be acquired within the first 45 min. Attenuation and decay-corrected images will be converted to standardized uptake value (SUV) maps through division by (injected activity per patient weight). The maximum SUV values over regions of interest will be determined for 10-min static images starting 35 min after the injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients will undergo standard-of-care investigations (CT imaging of adrenals and AVS) and the research test (11C-metomidate PET-CT) with a dose of 150 - 300 Megabecquerel (MBq) (11C-metomidate) to identify functional unilateral adrenal disease.
  Interventions: Combination Product: 11C-Metomidate PET/CT Scan

INTERVENTIONS:
Combination Product: 11C-Metomidate PET/CT Scan — 11C-Metomidate PET/CT imaging at Clinical Imaging Research Centre

SUMMARY:
10% of patients with hypertension potentially have the treatable condition - primary aldosteronism. Primary aldosteronism (PA) is caused by either bilateral adrenal disease (~40%), managed with lifelong medications; or unilateral disease (~60%), cured with laparoscopic surgery (adrenalectomy). Unfortunately, many patients with curable hypertension remain undiagnosed and consequently develop cardiac disease and strokes. The difficulty with identifying curable unilateral disease is due to adrenal vein sampling (AVS): an invasive, and technically-difficult procedure, with inconclusive results in 50% of patients. An alternative novel imaging, 11C-metomidate Positron emission tomography-computed tomography (PET-CT), can detect adrenal tumors, and concurrently confirm their over-activity. It is non-invasive, non-operator-dependent, and can identify more patients with curable hypertension.

Investigators hypothesize that 11C-metomidate PET-CT can accurately identify patients with surgically-curable unilateral adrenal disease among hypertensive Asians with primary aldosteronism.

DETAILED DESCRIPTION:
25 patients with confirmed PA who are keen for a surgical cure if unilateral PA is confirmed, will undergo conventional tests, CT, AVS, as well as 11C-metomidate PET/CT.

Results will be reviewed and discussed at a multidisciplinary meeting, and patients with unilateral PA will be offered surgery. Patients will be reviewed 6 months post surgery to assess for cure of PA.

ELIGIBILITY:
Inclusion Criteria:

• Primary aldosteronism, as defined in Endocrine Society Guidelines 2016, with positive confirmatory test (post-salt loading aldosterone >140pmol/L); or hypokalemia with undetectable renin levels and aldosterone >550pmol/L.

Exclusion Criteria:

* Inability to provide written informed consent
* < 21 years or > 70 years
* Chronic renal failure of Stage 3b or greater severity
* Severe or terminal medical condition(s)
* Contraindications to isotope scanning or CT Scan
* Contraindication to ingestion of corticosteroids

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Cure of Primary Aldosteronism Post-Adrenalectomy | 6 months
  Percentage of patients accurately identified with unilateral PA (determined by post-surgery biochemical cure) using 11C-metomidate PET/CT compared to percentage of patients accurately identified with unilateral PA (determined by post-surgery biochemical cure) using AVS

SECONDARY OUTCOMES:
Clinical Diagnosis of Unilateral Primary Aldosteronism | 6 months
  Percentage of patients accurately identified with unilateral PA (determined by clinical diagnosis made by multidisciplinary team) using 11C-metomidate PET/CT compared to percentage of patients accurately identified with unilateral PA (determined by clinical diagnosis made by multidisciplinary team) using AVS
Cost-Effectiveness of Diagnostic Test | 6 months
  Cost-Effectiveness of Diagnostic Test to identify unilateral PA

OTHER OUTCOMES:
Diagnostic criteria using 11C-Metomidate PET/CT | 6 months
  To assess the cut-off level of SUVmax which offers the best sensitivity and specificity for lateralisation in 11C-metomidate PET-CT

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puar TH, Khoo CM, Tan CJ, Tong AKT, Tan MCS, Teo AE, Ng KS, Wong KM, Reilhac A, O'Doherty J, Gomez-Sanchez CE, Kek PC, Yee S, Tan AWK, Chuah MB, Lee DHM, Wang KW, Zheng CQ, Shi L, Robins EG, Foo RSY; for the PA CURE investigators. 11C-Metomidate PET-CT versus adrenal vein sampling to subtype primary aldosteronism: a prospective clinical trial. J Hypertens. 2022 Jun 1;40(6):1179-1188. doi: 10.1097/HJH.0000000000003132. PMID 35703880